CLINICAL TRIAL: NCT07219680
Title: Intervention to Promote Communication Quality of Life for Persons With Language-Led Dementia and Their Partners: A Randomized Pilot Trial
Brief Title: Intervention for Communication Quality of Life in Primary Progressive Aphasia
Acronym: Multi-PA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R61AG089318 (NIH)
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Primary Progressive Aphasia(PPA); Semantic Dementia; Logopenic Progressive Aphasia (LPA); Nonfluent Aphasia, Progressive; Progressive Aphasia; Semantic Variant Primary Progressive Aphasia (svPPA); Semantic Aphasia; Logopenic Variant Primary Progressive Aphasia; Logopenic Variant of Primary Progressive Aphasia (LPA); Logopenic Progressive Aphasia; Nonfluent Variant Primary Progressive Aphasia (nfvPPA); Nonfluent Progressive Aphasia
Keywords: speech-language pathology; neurodegenerative disease; logopenic; nonfluent; semantic; script training; teletherapy; remote; multimodal communication training; partner training; augmentative and alternative communication; AAC; Communication Book; bilingual; Spanish; Hispanic; Latino
MeSH Terms: conditions — Aphasia, Primary Progressive; Frontotemporal Dementia; Primary Progressive Nonfluent Aphasia; Aphasia; Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: Participants in Arm 1, the immediate treatment group, will proceed immediately to initial assessments followed by the treatment phase (co-development of training materials and Multi-VISTA or Multi-LRT treatment).
  Participants in Arm 2, the waitlist control group, will undergo initial assessment followed by a waiting interval of 10 (Multi-VISTA) or 12 (Multi-LRT) weeks. Following the waiting period, they will be reassessed for cognitive-linguistic and participant-reported outcome measures prior to the treatment phase (co-development of training materials and Multi-VISTA or Multi-LRT treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Control (Other): Individuals in the waitlist-control group will undergo initial assessment followed by a waiting interval of 10 (Multi-VISTA) or 12 (Multi-LRT) weeks. Following the waiting period, they will again complete baseline assessments prior to the treatment phase (co-development of training materials and Multi-VISTA or Multi-LRT treatment).
  Interventions: Behavioral: Multicomponent Lexical Retrieval Training; Behavioral: Multicomponent Video Implemented Script Training in Aphasia
- Immediate Treatment (Experimental): Individuals in the immediate treatment group will undergo initial assessment followed immediately by the treatment phase (co-development of training materials and Multi-VISTA or Multi-LRT treatment).
  Interventions: Behavioral: Multicomponent Lexical Retrieval Training; Behavioral: Multicomponent Video Implemented Script Training in Aphasia

INTERVENTIONS:
Behavioral: Multicomponent Lexical Retrieval Training — In person or via teletherapy: A multi-component treatment incorporating elements of restitutive, compensatory, and care-partner focused interventions. Participants work on producing names of personally relevant target in multiple communication modalities. Biweekly (approximately one hour each) sessions with a clinician target multimodal communication and the use of strategies to support word retrieval. These skills are also trained via daily independent practice. The participant meets four times during the course of treatment with a study partner (e.g., spouse) for communication counseling, education, and practice of communication strategies.
  Other Names: Multi-LRT
Behavioral: Multicomponent Video Implemented Script Training in Aphasia — In person or via teletherapy: A multi-component treatment incorporating elements of restitutive, compensatory, and care-partner focused interventions. Treatment focuses on production of individually-tailored, personally relevant scripts. The participant completes 30 minutes per day of independent practice, during which they speak in unison with a video model. Biweekly (approximately one hour each) sessions with a clinician target clear and accurate script production, memorization, and conversational usage, as well as multimodal communication. The participant meets 6 times during the course of treatment with a study partner (e.g., spouse) for communication counseling, education, and practice of communication strategies.
  Other Names: Multi-VISTA

SUMMARY:
The goal of this clinical trial is to determine whether individually tailored speech-language telerehabilitation helps improve communication in people with primary progressive aphasia (PPA), a form of dementia that affects speech and language. The study will be offered to individuals who speak English and/or Spanish. The study will also document how acceptable and beneficial the program is to both patients and their care partners.

The main questions the study aims to answer are:

1. Is the telerehabilitation program feasible and acceptable for people with PPA and their care partners?
2. Do participants with PPA and care partners find treatment beneficial?
3. Which outcome measures are most useful for evaluating changes in communication and quality of life?
4. What patterns of treatment response are seen in participants after completing the program?

The program includes both speech-language therapy and training for care partners.

Participants with PPA will:

1. Complete virtual communication tasks and questionnaires before and after the program
2. Take part in online speech-language therapy sessions
3. Include their care partners in some parts of the program for training and support

ELIGIBILITY:
Inclusion Criteria for Persons with PPA:

* A PPA (Gorno-Tempini et al., 2011) or "PPA-plus" (Mesulam et al., 2001) diagnosis
* MMSE score of > 15 and must be able to produce single monosyllabic words intelligibly.
* Must speak English, Spanish or both languages (i.e., bilingual speakers of English or Spanish)
* Hearing and vision adequate for participation in teleconference meetings
* Must have a care partner available (someone who will commit to attending teleconference sessions weekly during treatment phases)

Inclusion criteria for Care Partners:

* Partners must express willingness to attend and participate in treatment sessions including those targeting dyadic communication goals
* Partners must speak English, Spanish or both languages (i.e., bilingual speakers of English or Spanish)
* Partner's hearing and vision should be adequate for participation in teleconference meetings

Exclusion criteria for persons with PPA:

* Other central nervous system or medical diagnosis that can account for symptoms
* Psychiatric diagnosis that can account for symptoms
* The participant and/or study partner must have basic experience using a computer.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-03 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in spoken naming of trained/untrained items | change from pre-treatment to post-treatment (11 weeks after treatment onset) and follow-up at 3 months post-treatment
  Percent correctly named trained/untrained pictures
Change in script production accuracy | change from pre-treatment to post-treatment (9 weeks after treatment onset) and follow-up at 3 months post-treatment
  Percent correct intelligible, scripted words for trained/untrained scripts
Change in barriers and facilitators in dyad conversation | change from pre-treatment to post-treatment (9-11 weeks after treatment onset) and follow-ups at 3 months post-treatment
  Number of conversation barriers and facilitators observed in conversation
Goal Attainment Score | change from pre-treatment to post-treatment (approximately 9-11 weeks after treatment onset) and follow-ups at 3 months post-treatment
  The Goal Attainment Score measures self-reported progress on personalized goals based on a five point scale, with higher values indicating better goal attainment. The minimum score is -2 (much less than expected) and the maximum score is +2 (much more than expected).

SECONDARY OUTCOMES:
Change on Quick Aphasia Battery | change from pre-treatment to post-treatment (approximately 9-11 weeks after treatment onset) and follow-ups at 3 months post-treatment
  The Quick Aphasia Battery is a standardized aphasia assessment.
Change on Aphasia Impact Questionnaire | change from pre-treatment to post-treatment (approximately 9-11 weeks after treatment onset) and follow-ups at 3 months post-treatment
  The Aphasia Impact Questionnaire is a psychosocial questionnaire for individuals with aphasia. Scores range from 0-84, with higher scores indicating greater impact of aphasia.
Acceptability and Perception of Change Survey | post-treatment (approximately 9-11 weeks after treatment onset)
  The Acceptability and Perception of Change Survey characterizes perceived response to treatment.
Change on Adult Carers Quality of Life Questionnaire | change from pre-treatment to post-treatment (approximately 9-11 weeks after treatment onset) and follow-ups at 3 months post-treatment
  The Adult Carers Quality of Life Questionnaire is a measure evaluating quality of life for caregivers. Scores range from 0-100, with higher scores indicating greater quality of life.
Change on Brief - Coping Orientation to Problems Experienced Inventory (Brief-COPE) | change from pre-treatment to post-treatment (approximately 9-11 weeks after treatment onset) and follow-ups at 3 months post-treatment
  The Brief-COPE is a survey characterizing care partner use of coping strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Maya L Henry, PhD, Principal Investigator — University of Texas at Austin; Stephanie M Grasso, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Because of the possibility of deductive disclosure of subjects with unusual characteristics and the sensitive nature of the protected health information obtained in this trial, we will make decisions about data sharing on request, with IRB oversight.

REFERENCES:
- [Background] Henry ML, Hubbard HI, Grasso SM, Mandelli ML, Wilson SM, Sathishkumar MT, Fridriksson J, Daigle W, Boxer AL, Miller BL, Gorno-Tempini ML. Retraining speech production and fluency in non-fluent/agrammatic primary progressive aphasia. Brain. 2018 Jun 1;141(6):1799-1814. doi: 10.1093/brain/awy101. PMID 29718131
- [Background] Henry ML, Hubbard HI, Grasso SM, Dial HR, Beeson PM, Miller BL, Gorno-Tempini ML. Treatment for Word Retrieval in Semantic and Logopenic Variants of Primary Progressive Aphasia: Immediate and Long-Term Outcomes. J Speech Lang Hear Res. 2019 Aug 15;62(8):2723-2749. doi: 10.1044/2018_JSLHR-L-18-0144. Epub 2019 Aug 7. PMID 31390290
- [Background] Dial HR, Hinshelwood HA, Grasso SM, Hubbard HI, Gorno-Tempini ML, Henry ML. Investigating the utility of teletherapy in individuals with primary progressive aphasia. Clin Interv Aging. 2019 Feb 25;14:453-471. doi: 10.2147/CIA.S178878. eCollection 2019. PMID 30880927
- See also: University of Texas Aphasia Research and Treatment Lab — https://slhs.utexas.edu/research/aphasia-research-treatment-lab
- See also: University of Texas Aphasia Multilingual Aphasia and Dementia Research Lab — https://slhs.utexas.edu/research/multilingual-aphasia-and-dementia-research-lab/about-lab